CLINICAL TRIAL: NCT04320459
Title: Alexithymia in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Other Study IDs: MedeniyetRomato
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; alexithymia
MeSH Terms: conditions — Spondylitis, Ankylosing; Affective Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ankylosing spondylitis: 55 patients having Ankylosing Spondylitis (AS) for at least 1 year diagnosed according to the ASAS classification criteria who presented to our hospital's outpatient clinic
  Interventions: Diagnostic Test: Bath Ankylosing Spondylitis Metrology Index (BASMI); Diagnostic Test: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI); Diagnostic Test: Bath Ankylosing Spondylitis Functional Index (BASFI); Diagnostic Test: Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL); Diagnostic Test: Toronto Alexithymia Scale-20 (TAS-20); Diagnostic Test: Beck's Depression Inventory (BDI)
- healthy control: age and sex matched healthy controls
  Interventions: Diagnostic Test: Bath Ankylosing Spondylitis Metrology Index (BASMI); Diagnostic Test: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI); Diagnostic Test: Bath Ankylosing Spondylitis Functional Index (BASFI); Diagnostic Test: Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL); Diagnostic Test: Toronto Alexithymia Scale-20 (TAS-20); Diagnostic Test: Beck's Depression Inventory (BDI)

INTERVENTIONS:
Diagnostic Test: Bath Ankylosing Spondylitis Metrology Index (BASMI) — It characterises the spinal mobility of patients with ankylosing spondylitis. Cervical rotation, tragus-wall distance, lateral lumbar flexion, anterior lumbar flexion (modified schober), intermalleolar distance were measured. The total score of the 5 measurements was taken, the score range was 0-10, the low score meant that the spinal movement was better.
Diagnostic Test: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) — It assess the disease activity. It was evaluated with a 6-question questionnaire. After taking the answer of each question out of 10, the total of the points was calculated by dividing the number of questions.
Diagnostic Test: Bath Ankylosing Spondylitis Functional Index (BASFI) — It assess functional status. It was evaluated with a 10-question questionnaire. After taking the answer of each question out of 10, the total of the points was calculated by dividing the number of questions.
Diagnostic Test: Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) — It evaluates quality of life. Each statement on the ASQoL (18-item) is given a score of "1" or "0". A score of "1" is given where the item is affirmed, indicating adverse QoL. All item scores are summed to give a total score or index. Scores can range from 0 (good QoL) to 18 (poor QoL).
Diagnostic Test: Toronto Alexithymia Scale-20 (TAS-20) — It assess alexithymia. It is a 20 item questionnaire and each item is evaluated in a Likert type scale with five intervals (1= strongly disagree, 5=strongly agree). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.
Diagnostic Test: Beck's Depression Inventory (BDI) — It assess depression status. It is a 21-question multiple-choice self-report inventory, each set is ranked in terms of severity and scored from 0 to 3 with a total summed score range of 0-63. Higher scores indicate greater depressive severity. Conventional cutoffs are 0-9 for normal range, 10-18 for mild to moderate depression, 19-29 for moderate to severe depression, and 30-63 for severe depression.

SUMMARY:
The study included 55 patients having Ankylosing Spondylitis (AS) for at least 1 year diagnosed according to the ASAS classification criteria who presented to our hospital's outpatient clinic and 55 healthy subjects. Demographic data were recorded for 55 AS patients who were subsequently assessed using the BASMI (Bath Ankylosing Spondylitis Metrology Index) in terms of elasticity and spinal mobility as well as the BASFI (Bath Ankylosing Spondylitis Functional Index) to determine functional status, the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) to assess the disease activity and the ASQoL (Ankylosing Spondylitis Quality of Life Questionnaire) to evaluate quality of life. The Toronto Alexithymia Scale-20 (TAS-20) was used for assessment of alexithymia and Beck's Depression Inventory (BDI) for depression among patients.

DETAILED DESCRIPTION:
The study included 55 patients having Ankylosing Spondylitis (AS) for at least 1 year diagnosed according to the ASAS classification criteria who presented to our hospital's outpatient clinic and 55 healthy subjects. Demographic data were recorded for 55 AS patients who were subsequently assessed using the BASMI (Bath Ankylosing Spondylitis Metrology Index) in terms of elasticity and spinal mobility as well as the BASFI (Bath Ankylosing Spondylitis Functional Index) to determine functional status, the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) to assess the disease activity and the ASQoL (Ankylosing Spondylitis Quality of Life Questionnaire) to evaluate quality of life. The Toronto Alexithymia Scale-20 (TAS-20) was used for assessment of alexithymia and Beck's Depression Inventory (BDI) for depression among patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as AS for at least 1 year according to the ASAS classification criteria
* over 18 years old

Exclusion Criteria:

* fibromyalgia
* age less than 18 years
* vision and hearing impairment
* neurological disease (Parkinson's disease, multiple sclerosis, cerebrovascular disease),
* history of a psychiatric disorder (schizophrenia, bipolar disorder)
* history of chronic condition (DM, thyroid disease) or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study included 55 patients having AS for at least 1 year diagnosed according to the ASAS classification criteria who presented to our hospital's outpatient clinic and 55 healthy subjects.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Alexithymia rate in AS patients and controls according to Toronto Alexithymia Scale-20 | 7 months
Depression rate in AS patients and controls according to Beck Depression Inventory | 7 months
Relationship between alexithymia and depression and functional indexes (BASFI, BASMI, BASDAI, ASQoL) | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided